CLINICAL TRIAL: NCT00557817
Title: Darbepoetin-alpha and i.v. Iron Administration After Autologous Hematopoietic Stem Cell Transplantation : a Prospective Randomized Trial
Brief Title: Erythropoietin (Epo) and Venofer Trial After Autologous Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Amgen (Industry); KU Leuven (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Beguin Yves, University Hospital of liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJE0301
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2008-08

CONDITIONS: Hematological Malignancies
Keywords: HCT; autologous; erythropoiesis; iron saccharate; erythropoietin; darbepoetin alpha
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Darbepoetin alfa; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): No medication given
- 2 (Active Comparator): Aranesp 300 µg/15 days
  Interventions: Drug: Darbepoetin alpha (Aranesp)
- 3 (Active Comparator): Aranesp 300 µg/15 days. Venofer 200 mg on days 28, 42, and 56 after the transplant.
  Interventions: Drug: Darbepoetin alpha (Aranesp); Drug: Iron saccharate (Venofer)

INTERVENTIONS:
Drug: Darbepoetin alpha (Aranesp) — Darbepoetin alpha (Aranesp) will be administered subcutaneously (s.c.) at the dose of 300 µg. The first dose will be given on day 28 and the following doses at 2-week intervals around days 42, 56, 70, 84, 98 and 112 post-transplant. Once the target Hb (13 g/dL) has been attained, the dose of Aranesp will be reduced by half to 150 µg. If the Hb increases to > 14 g/dL, Aranesp will be withheld and resumed at the dose of 150 µg when the Hb decreases < 13 g/dL. If the Hb decreases to < 12 g/dL, the dose of Aranesp will be increased to 300 µg again.
  Other Names: Aranesp
  Arms: 2; 3
Drug: Iron saccharate (Venofer) — Iron saccharate (Venofer) will be administered intravenously (i.v.) at the dose of 200 mg (2 vials of Venofer) on days 28, 42 and 56 after the transplant. Venofer will be diluted in 250 ml saline and infused over 60 minutes. Iron will be omitted in patients with severe iron overload (serum ferritin > 2500 µg/L in the absence of inflammation or liver necrosis) or elevated transferrin saturation (TS > 60%) between days 21 and 56. No iron supplementation will be allowed in arm 1. No iron supplementation will be allowed in arm 2 before day 70 after the transplant. In arms 2 and 3, if patients have evidence of functional iron deficiency (transferrin saturation < 20%) on day 70 or later, they will receive 300 mg of Venofer over 90 min, for a minimum of 2 doses.
  Other Names: Venofer
  Arms: 3

SUMMARY:
Darbepoetin-alpha and i.v. iron administration after autologous hematopoietic stem cell transplantation for hematological malignancies : a prospective randomized trial.

DETAILED DESCRIPTION:
1. Outline:

   A 3-arm prospective randomized study of darbepoetin alpha administration after autologous PBSC transplantation. Patients in the first arm will receive neither darbepoetin alpha nor i.v. iron. Patients in the second arm will receive darbepoetin alpha (Aranesp) alone starting on day 28 after the transplant. Patients in the third arm will receive darbepoetin alpha (Aranesp) and i.v. iron saccharate (Venofer). The plan is to include 25 patients in each arm.

   In September 2006, all 75 planned patients have been included. Whereas preliminary analysis shows that Aranesp therapy significantly improves Hb recovery after autologous PBSC transplantation, the additional impact of Venofer therapy remains statistically not significant. However, this is a very important point, because Venofer therapy could potentially improve response and decrease the overall cost of treatment. Therefore, to increase the statistical power of the study, 50 additional patients will be included. Randomisation will now become limited to arms 2 (Aranesp) and 3 (Aranesp + Venofer).
2. Randomization:

   Patients will be randomized 1:1:1 between the "Control", "Aranesp alone" and "Aranesp + Venofer" arms. Randomization will be carried out following a computer-generated randomization list blinded for personnel involved in clinical care of the patients.

   Randomization will be carried out centrally in Liège by faxing the inclusion form at the following number : 32-4-3668855. This should be done around day 21 post-transplant.

   Starting in September 2006, patients will be randomized 1:1 between the "Aranesp alone" and "Aranesp + Venofer" arms, using a computer-generated randomization list.
3. Study drug administration:

   * Darbepoetin alpha administration : Darbepoetin alpha (Aranesp) will be administered s.c. at the dose of 300 µg. The first dose will be given on day 28 and the following doses at 2-wk intervals around days 42, 56, 70, 84, 98, and 112 post-transplant. Once the target Hb (13 g/dL) has been attained, the dose of Aranesp will be reduced by half to 150 µg. If the Hb increases to > 14 g/dL, Aranesp will be withheld and resumed at the dose of 150 µg when the Hb decreases < 13 g/dL. If the Hb decreases to < 12 g/dL, the dose of Aranesp will be increased to 300 µg again.
   * Iron administration: Iron saccharate (Venofer) will be administered i.v. at the dose of 200 mg (2 vials of Venofer) on days 28, 42, and 56 after the transplant. Venofer will be diluted in 250 ml saline and infused over 60 minutes. Iron will be omitted in patients with severe iron overload (serum ferritin > 2500 µg/L in the absence of inflammation or liver necrosis) or elevated transferrin saturation (TS > 60%) between days 21 and 56. No iron supplementation will be allowed in arm 1. No iron supplementation will be allowed in arm 2 before day 70 after the transplant. In arms 2 and 3, if patients have evidence of functional iron deficiency (Transferrin saturation < 20%) on day 70 or later, they may receive 300 mg of Venofer over 90 min, for a minimum of 2 doses.
4. Transfusions:

   One red blood cell (RBC) unit will be transfused if Hb value is between 7.0 and 7.9 g/dL. Two RBC units will be transfused if Hb value is below 7 g/dL. Platelets will be transfused if needed, as per the institution's standards.
5. Follow-up:

   * Clinical follow-up : Potential toxicities associated with Aranesp or Venofer will be carefully monitored per the institution's standards. Blood pressure will be recorded around days 28, 42, 56, 70, 84, 98, 112, and 126 after the transplant. Serious adverse events (such as infections, bleeding, disease progression, any hospitalization) will be recorded. In case of serious adverse event judged as potentially related to Aranesp or Venofer, the principal investigator will be immediately notified so as to jointly decide on possible discontinuation of either drug.

   Quality-of-life (QOL) evaluations will be carried out at baseline (day 28) as well as on days 70 and 126 after the transplant, i.e. after 3 and 7 doses of Aranesp therapy. This will be accomplished by providing the patient will the validated FACT-anemia questionnaire. The questionnaire will be filled out by the patient and returned to the principal investigator.
   * Laboratory analyses: Complete blood counts will be determined in an automated cell counter. Percentage and absolute reticulocyte count will be obtained locally by an automated cytofluorometric method. Serum erythropoietin (Epo) levels will be measured centrally in Liège on stored samples by a commercially available radioimmunoassay (Incstar Corp., Stillwater, MN, USA). Based on regression equations obtained in appropriate reference subjects between Hct on the one hand and log (Epo) on the other, predicted log (Epo) values are derived for each Hct and O/P ratios of observed/predicted Epo values will be calculated. Serum soluble transferrin receptor (sTfR), a quantitative measure of total erythropoietic activity, will be measured centrally in Liège on stored samples by a commercially available ELISA (R&D, Minneapolis, MN, USA). Normal values range from 3,000 to 7,000 µg/L. Serum iron, transferrin saturation and ferritin, as well as standard biochemical values, will be measured locally by standard methods.

   On days 28 and 42, 5 ml of blood without anticoagulant will be collected and centrifuged within 2 hours, serum will be separated and 2 ml of serum will be stored at -28°C. Stored samples will be collected by the local investigator and finally stored in Liège. Serum Epo and soluble TfR will be assayed later on all samples simultaneously.
6. Data collection and analysis:

Data will be collected at each center on protocol forms. The coordinating data manager from Liège will verify the completeness and accuracy of data collected. The coordinating data manager will be responsible for entering these data into the central database. All statistical analyses will be performed centrally in Liège.

ELIGIBILITY:
Inclusion criteria:

* Male or female; female patients must use a reliable contraception method
* Age > 16 yrs and < 70 yrs
* No terminal organ failure
* Written informed consent given by patient or his/her guardian if of minor age.
* Adequate iron stores (serum ferritin > 100 µg/L) on day 21 post-transplant.
* Adequate marrow recovery, as shown by: neutrophils > 1,000/µL, platelet transfusion independence
* PBSC (not marrow) transplantation

Exclusion criteria:

* HIV positive
* Known allergy to recombinant human erythropoietin or i.v. iron saccharate
* Evidence of active hemorrhage, hemolysis, vitamin B12 or folate deficiency on day 28 post-transplant (inclusion into the protocol may then be delayed up until day 42 if the problem is resolved)
* Uncontrolled infection, arrythmia or hypertension on day 28 post-transplant (inclusion into the protocol may then be delayed up until day 42 if the problem is resolved)
* Evidence of severe iron overload (transferrin saturation > 60%, serum ferritin > 2500 µg/L on day 21 post-transplant)

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Median time to achieve hemoglobin (Hb) level > 13 g/dL in each arm. | 126 days after hematocrit (HCT)
Proportion of complete correctors (i.e. patients reaching Hb > 13 g/dL) before day 126 in each arm. | 126 days after HCT

SECONDARY OUTCOMES:
Median time to increase Hb level by > 2 g/dL in each arm. | 126 days after HCT
Proportion of responders (i.e. patients increasing Hb by > 2 g/dL) before day 126 in each arm. | 126 days after HCT
Proportion of correctors (i.e. patients reaching Hb > 12 g/dL) before day 126 in each arm. | 126 days after HCT
Proportion of patients requiring red blood cell transfusions between day 28 and day 126 in each arm. | 126 days after HCT
Total number of red blood cell transfusions between day 28 and day 126 in each arm. | 126 days after HCT
Area under the curve of mean Hb level between day 28 and day 126 after the transplant in each arm. | 126 days after HCT
Mean Hb values on days 42, 56, 70, 84, 98, 112, and 126 in each arm. | 126 days after HCT
Mean change in Quality Of Life (QOL) measurements between day 28 and day 126 in each arm. | 126 days after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Study Chair — CHU-ULg; Frederic Baron, MD, PhD, Principal Investigator — CHU-ULg; Johan Maertens, MD, PhD, Principal Investigator — KU Leuven; Rik Schots, MD, Principal Investigator — Vrije Universiteit Brussel; Bernard DePrijck, MD, Principal Investigator — CHR Citadelle
Locations (4):
- Belgium (4):
  - Vrije Universiteit Brussel, Brussels, Brussels Capital
  - Katholieke Universiteit Leuven, Leuven, Leuven
  - CHR la citadelle, Liège, Liege
  - CHU Sart Tilman, Liège, Liege